CLINICAL TRIAL: NCT01840696
Title: Regional and Global Left Ventricular Mechanical Dyssynchrony in the Diagnosis of Obstructive Coronary Artery Disease on Rest and Regadenoson Stress Rubidium Myocardial Perfusion PET
Brief Title: Phase Analysis and Obstructive CAD on Rubidium PET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI leaving facility
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Fabio Esteves, MD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00062632; REGA12I11 (Other: Other)
Record Dates: First submitted 2013-04-16; First posted 2013-04-26 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regadenoson (Experimental)
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Vasodilator stress testing
  Other Names: Lexiscan

SUMMARY:
Rubidium myocardial perfusion PET is an imaging test used to diagnose patients with abnormal blood flow to the heart secondary to narrowing of the heart vessels.

Phase analysis is a computer method that is applied after the PET test is done. It is used to determine when a region of the heart contracts relative to other heart regions in the heart beating cycle. Initial data suggest that regions of the heart with abnormal blood flow change the pattern of contraction from rest to stress conditions. That is, regions of the heart with abnormal blood supply become dyssynchronous when compared to the normal regions of the heart.

This study will investigate whether phase analysis may aid the visual interpretation of rubidium myocardial perfusion PET studies by determining the areas of the heart that are not beating in synchrony with the normal heart regions. This information will be used as a proxy for poor blood supply. The gold standard will be coronary angiography by which the percent narrowing of the heart vessels is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* referred for myocardial perfusion imaging for suspected obstructive CAD
* 18 years of age or older.

Exclusion Criteria:

* Contraindications to regadenoson radionuclide imaging including severe reactive airway disease, unstable crescendo angina, high grade AV block, caffeine within 24 hours
* Documented prior myocardial infarction
* Severe claustrophobia
* Patients who may be pregnant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Stress/rest differences in global left ventricular mechanical contraction bandwidth. | Up to 12 months
  The investigators will measure the percent change in global left ventricular mechanical contraction bandwidth between stress and rest perfusion imaging as measured by phase analysis.
  Two patients were enrolled but the data were not analyzed.

SECONDARY OUTCOMES:
Stress/rest differences in segmental left ventricular mechanical contraction bandwidth. | Up to 12 months
  The investigators will measure the percent change in segmental (each of 3 major coronary arteries) left ventricular mechanical contraction bandwidth between stress and rest perfusion imaging as measured by phase analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Esteves, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States